CLINICAL TRIAL: NCT06723054
Title: Prevention and Arrest of Root Caries Lesions with High Fluoride Concentration Mouthwash Versus Normal Fluoride Concentration Mouthwash in Elderly Patients: a Randomized, Double-blind Controlled Trial.
Brief Title: Prevention and Arrest of Root Caries Lesions with High Fluoride Concentration Mouthwash Versus Normal Fluoride Concentration Mouthwash in Elderly Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murali Srinivasan, Dr. med. dent., BDS, MDS, MBA, MAS (Other)
Responsible Party: Sponsor-Investigator, Murali Srinivasan, Dr. med. dent., BDS, MDS, MBA, MAS, Prof. Dr. med. dent., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UZH_ABS_2021_9; UZH_ABS_2021_9 (Other: University Zurich, ZZM / ABS)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Root Caries
Keywords: Elders; Root caries lesions; Prevention; Mouthwash
MeSH Terms: conditions — Root Caries | interventions — Erythritol

STUDY DESIGN:
Intervention Model Description: This study is designed to be a double-blind, randomized, controlled, parallel, single-center, intention-to treat (ITT), trial with an allocation ratio of 1: 1: 1 and of a non-inferiority framework. The participants will be randomly allotted to one of the three study groups.
Who Masked: Participant, Investigator
Masking Description: The participants and the investigators will be blinded to the randomization sequence as well as the prevention group. They will both not be aware of which mouthwash was used by the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (CG) (Placebo Comparator): Regular fluoride 220 ppm F mouthwash without erythritol
  Interventions: Other: regular fluoride 220 ppm F mouthwash without erythritol
- Intervention group #1 (IG1) (Active Comparator): 220 ppm F mouthwash with erythritol
  Interventions: Other: regular fluoride 220 ppm F mouthwash with erythritol
- Intervention group #2 (IG2) (Active Comparator): 500 ppm F mouthwash with erythritol
  Interventions: Other: high fluoride 500 ppm F mouthwash with erythritol

INTERVENTIONS:
Other: regular fluoride 220 ppm F mouthwash without erythritol — The participants will be asked to rinse once daily with a regular fluoride 220 ppm F mouthwash without erythritol.
  Arms: Control group (CG)
Other: regular fluoride 220 ppm F mouthwash with erythritol — The participants will be asked to rinse once daily with a regular fluoride 220 ppm F mouthwash with erythritol.
  Arms: Intervention group #1 (IG1)
Other: high fluoride 500 ppm F mouthwash with erythritol — The participants will be asked to rinse once daily with a high fluoride 500 ppm F mouthwash with erythritol.
  Arms: Intervention group #2 (IG2)

SUMMARY:
The study evaluats the effectiveness of regular fluoride 220 ppm F with erythritol and high fluoride 500 ppm F with erythritol mouthwashes against a placebo (regular fluoride 220 ppm F mouthwash) in the prevention of new root caries lesions.

DETAILED DESCRIPTION:
Preserving natural teeth becomes essential to avoid complex restorative procedures in old age. For this the concepts of preventive treatment constitute an important point. The method of topical application via fluorides is a widely used and well-known technique for prevention of caries. Numerous studies have demonstrated the preventive effect of fluorides on caries. The prevention of root caries and the effectiveness of fluorides will depend mainly on two factors used: first is the fluoride agent, and the second is fluoride content. There is abundant evidence with regard to the preventive effect of high fluoride applications on the root caries. Furthermore, it has also been recommended on the regular use of high fluoride 5000 ppm F toothpaste twice daily in the prevention and inactivating the root caries in adults. However, high fluoride toothpastes are fairly expensive and not available as over-the-counter (OTC) products and require a prescription. This may be an aspect when the elders have limited access. A more economical solution and one which can be easily procured is deemed necessary.

Mouth rinses are considered as cosmetic products and are available as OTC products and do not require prescriptions. They are also relatively less expensive in comparison to the high fluoride toothpastes. Fluoridated mouthwashes are generally recommended in moderate-high caries risk population or individual. The normal fluoride range in a mouth wash is normally between 100 ppm to 500 ppm F. This may not be sufficient to bring a preventive effect in high risk individuals. It has been demonstrated that a small positive trend for sodium fluoride (NaF) mouth rinses against placebo in reducing the initiation of coronal and root caries.

Erythritol is a natural sugar substitute and is frequently used as a sweetener. It is easily excreted by the kidneys and does not increase the blood sugar. It is often an additive in mouthwashes as a sweetening agent. It is known to have anti-plaque aggregating and bacteriostatic effect.

Perhaps, the use of erythritol in regular fluoride mouthwash (220 ppm F) in combination with high F mouthwash (500 ppm F) might be beneficial and augment the preventive effect of fluoride in mouth rinses. This may be a viable alternative to expensive and prescription options.

Therefore, the primary objective of this study is to evaluate the effectiveness of regular fluoride 220 ppm F with erythritol and high fluoride 500 ppm F with erythritol mouthwashes against a placebo (regular fluoride 220 ppm F mouthwash) in the prevention of new root caries lesions.

The secondary endpoints/outcome set for this study is the number of arrested root surface caries after intervention with the test products (i.e., a change of root surface caries from ICDAS classification 1 to 2 and 3 to 4, respectively will be considered as arresting).

The tertiary endpoint/outcome set for this study are as follows: 1. Incidence of new coronal caries after the intervention with the test products and 2. the number of arrested coronal caries after the intervention with the test products.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥60 years
* Dentinal root caries lesions with no painful symptomology
* Minimum of 3 teeth present in the mouth
* Can follow instructions for oral hygiene

Exclusion Criteria:

* Symptomatic carious teeth
* Root surface active lesion which is easily penetrated by sharp probe with light force (ICDAS Grade 3 and soft needs to be filled)
* Non-carious attrition, erosion or abrasion cavities
* Periodontally compromised teeth with Grade 3 mobility, and active signs of infections.
* Not willing or able to sign informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of new root surface caries (RCnew) on the exposed sound root surfaces | 180 days
  For this purpose of the trial each of the four tooth surfaces (i.e. distal, mesial, buccal, oral) will be assessed. All the exposed sound root surfaces will be taken into account and assessed at timepoints T0, T1 and T2 and will be compared to the tooth status at the previous visit. A new root surface caries is defined if a sound root surface, ICDAS 0, becomes a ICDAS 1, 2, 3, 4 or 6.

SECONDARY OUTCOMES:
Number of arrested root surface caries (RCarrested) on the exposed sound root surfaces | 180 days
  For this purpose of the trial each of the four tooth surfaces (i.e. distal, mesial, buccal, oral) will be assessed. All the active root surfaces caries which became a arrested root surfaces caries will be taken into account. The assessment will take place at timepoints T0, T1 and T2. The tooth status will each time be compared to the tooth status at the previous visit. A arrested root surface caries is defined if a active root surface caries lesion (ICDAS: 1 or 3) that becomes inactive root surface caries lesion (ICDAS: 2 or 4).

OTHER OUTCOMES:
1. Incidence of new active coronal caries (DCnew) and 2. Number of arrested coronal caries (DCarrested) | 180 days
  For the other Outcome 1. each of the five tooth surfaces (i.e. distal, mesial, buccal, oral, and occlusal) will be assessed. The tooth surfaces will be assessed at timepoints T0, T1 and T2 and will be compared to the tooth status at the previous visit. A new coronal caries (DCnew) is defined if a sound tooth surface, ICDAS 0, becomes a ICDAS 1, 2, 3, 4, 5 or 6. For the other Outcome 2. each of the five tooth surfaces (i.e. distal, mesial, buccal, oral, and occlusal) will be assessed. All the active coronal caries which became an arrested coronal caries will be taken into account. The assessment will take place at timepoints T0, T1 and T2. The tooth status will each time be compared to the tooth status at the previous visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Center for Dental Medicine, Clinic of General, Special care, and Geriatric Dentistry, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided